CLINICAL TRIAL: NCT06401720
Title: Respiratory Immune Responses in Human Influenza Virus Infection Across Age to Understand What Dictates Disease Severity
Brief Title: Age Related Differences in Respiratory Immune Responses in Influenza Virus Infection
Acronym: NPA-DC
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anna Smed Sörensen, Professor, Karolinska Institutet
Other Study IDs: 2023-01776
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Influenza A Infection; Influenza B Virus Infection; SARS CoV 2 Infection; RSV Infection
Keywords: Influenza A virus (IAV); Influenza B virus (IBV); SARS CoV 2; respiratory syncytial virus (RSV); immunology; age-related differences
MeSH Terms: conditions — COVID-19; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cryopreserved PBMCs. Plasma. Serum. Nasopharyngeal aspirate liquid. Endotracheal tube aspirate liquid. Nasal swab liquid. Nasopharyngeal swab liquid. Nasal curette liquid. Breath Explor devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with airway infection. Enrolled while seeking health care or when hospitalized.
- Controls: Subjects without airway infection.

SUMMARY:
The goal of this observational study is to understand immune responses to viral airway infection in adults, including the elderly. The main question(s) to answer is/are:

Why do some individuals acquire only asymptomatic or mild Influenza A virus (IAV) infection while others become severely ill and even succumb to the same disease?

Participants will be asked to donate samples when seeking health care for influenza-like symptoms or if hospitalized for IAV or SARS-CoV-2. Samples asked for are:

* Blood sample by venepuncture
* Blood sample by capillary sampling
* Nasopharyngeal aspirate
* Nasopharyngeal swab
* Endotracheal tube aspirate
* Nasal swab
* Nasal curette
* Breath Explor (sampling of expired air)

Researchers will compare obtained results with the same type of samples from healthy controls.

DETAILED DESCRIPTION:
This observational study will specifically investigate different immunological parameters in blood and at the site of infection in patients with IAV symptoms or confirmed infection to understand parameters related to disease course. Blood and airway samples will be analyzed for immune cell subsets and their functionality, antibodies and other soluble mediators and linked to clinical data. Immune cells will be analyzed using multi-color flow cytometry, RNA sequencing, and in vitro functionality assays. Fluids (plasma, serum, supernatants from airway samples and cell culture supernatants) will be analyzed using ELISA (and or similar methods), proximity extension assay (Olink), etc.

ELIGIBILITY:
Inclusion Criteria Patients:

* Influenza A like symptoms and/or
* Confirmed airway infection

Exclusion Criteria Patients:

* Current malignancies
* Immunosuppressive treatment, not including/except hydrocortisone

Exclusion Criteria Controls:

* Airway infection within the past four weeks
* Ongoing antibiotic treatment
* Immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are from primary care clinics, hospitalized, or household contacts of subjects seeking health care at a primary care clinic.
  The study population is included in the greater Stockholm area within the Region Stockholm health care region.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of immune cells | Samples are taken at several different occasions when the patient is experiencing an airway infection and during convalescence. Samples are taken during a time frame of up to 6 months.
  Flow cytometric analysis of white blood cell phenotype and frequency in PBMC, nasopharyngeal aspirate, nasopharyngeal swab, nasal swab, nasal curette, and endotracheal tube aspirate samples.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Smed Sörensen, PhD, Principal Investigator — Karolinska Institutet
Locations (5):
- Sweden (5):
  - Södertälje Sjukhus, Södertälje
  - Familjeläkarna, Stockholm
  - Haga Närakut, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Sabbatsbergs sjukhus, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu M, Charles A, Cagigi A, Christ W, Osterberg B, Falck-Jones S, Azizmohammadi L, Ahlberg E, Falck-Jones R, Svensson J, Nie M, Warnqvist A, Hellgren F, Lenart K, Arcoverde Cerveira R, Ols S, Lindgren G, Lin A, Maecker H, Bell M, Johansson N, Albert J, Sundling C, Czarnewski P, Klingstrom J, Farnert A, Lore K, Smed-Sorensen A. Delayed generation of functional virus-specific circulating T follicular helper cells correlates with severe COVID-19. Nat Commun. 2023 Apr 15;14(1):2164. doi: 10.1038/s41467-023-37835-9. PMID 37061513
- [Background] Vangeti S, Falck-Jones S, Yu M, Osterberg B, Liu S, Asghar M, Sonden K, Paterson C, Whitley P, Albert J, Johansson N, Farnert A, Smed-Sorensen A. Human influenza virus infection elicits distinct patterns of monocyte and dendritic cell mobilization in blood and the nasopharynx. Elife. 2023 Feb 8;12:e77345. doi: 10.7554/eLife.77345. PMID 36752598
- [Background] Cagigi A, Yu M, Osterberg B, Svensson J, Falck-Jones S, Vangeti S, Ahlberg E, Azizmohammadi L, Warnqvist A, Falck-Jones R, Gubisch PC, Odemis M, Ghafoor F, Eisele M, Lenart K, Bell M, Johansson N, Albert J, Salde J, Pettie DD, Murphy MP, Carter L, King NP, Ols S, Normark J, Ahlm C, Forsell MN, Farnert A, Lore K, Smed-Sorensen A. Airway antibodies emerge according to COVID-19 severity and wane rapidly but reappear after SARS-CoV-2 vaccination. JCI Insight. 2021 Nov 22;6(22):e151463. doi: 10.1172/jci.insight.151463. PMID 34665783
- [Background] Falck-Jones S, Vangeti S, Yu M, Falck-Jones R, Cagigi A, Badolati I, Osterberg B, Lautenbach MJ, Ahlberg E, Lin A, Lepzien R, Szurgot I, Lenart K, Hellgren F, Maecker H, Salde J, Albert J, Johansson N, Bell M, Lore K, Farnert A, Smed-Sorensen A. Functional monocytic myeloid-derived suppressor cells increase in blood but not airways and predict COVID-19 severity. J Clin Invest. 2021 Mar 15;131(6):e144734. doi: 10.1172/JCI144734. PMID 33492309
- See also: Home page of the research group performing the study — https://ki.se/en/research/groups/respiratory-and-systemic-immune-responses-in-human-pulmonary-viral-infection-and#tab-start